CLINICAL TRIAL: NCT05473962
Title: Mid-Term Follow-up Assessment After Exposure to Natural Disaster
Acronym: MFAE-ND
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 22-HPNCL-02
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-03

CONDITIONS: Psychiatric Disorder
Keywords: Post-traumatic stress disorder (PTSD)
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exposed to Alex storm: Child and/or young adult aged under 18 at the time of exposure having been assessed by the CUMPS teams during the "ALEX Storm" interventions of October 2020
  Interventions: Diagnostic Test: assessment and quantification of symptoms related to post-traumatic stress.

INTERVENTIONS:
Diagnostic Test: assessment and quantification of symptoms related to post-traumatic stress. — Semi-structured interview based on the Clinician-Administered PTSD scale for DSM-5 Child/Adolescent -CAPS-CA-5. This instrument allows for the This instrument is validated in English, and a French translation was carried out by the investigators (translation/back-translation method). The instrument uses the DSM-5 diagnostic criteria for post-traumatic stress disorder (PTSD).

SUMMARY:
The present study proposes to carry out an evaluation of the children of adolescents who were seen by the teams of the Cellules d'Urgence Médico-Psychologique (CUMP) following the Alex storm in October 2020. A clinical child psychiatric and psychological evaluation will be carried out, with collection of socio-demographic data

DETAILED DESCRIPTION:
Description: Assessment 24 months after exposure to a natural disaster of the clinical condition of children and adolescents cared for by medical-psychological emergency teams (CUMP) by measuring the frequency of clinical disorders and the intensity of symptoms and by comparing their clinical condition to that assessed immediately after exposure.

* Primary endpoint:

Semi-structured interview based on the Clinician-Administered PTSD scale for DSM-5 Child/Adolescent -CAPS-CA-5. This instrument allows for the assessment and quantification of symptoms related to post-traumatic stress. This instrument is validated in English, and a French translation was carried out by the investigators (translation/back-translation method). The instrument uses the DSM-5 diagnostic criteria for post-traumatic stress disorder (PTSD).

* Secondary endpoints:
* The intensity of the symptoms of this PTSD will be assessed by the Young Child PTSD checklist (YCPC) (Scheeringa, 2013; translation of the French version: Thümmler et al., 2017) for young children under the age of 7. For children over 7 years of age, it will be assessed by the Child PTSD checklist, child version (CPC) (Scheeringa, 2014; translation and validation of the French version: Gindt et al., 2020).
* Patient Health Questionnaire 13 items (PQH13). This simple and quick to use instrument allows a systematic assessment of somatization in children. This questionnaire will be offered to parents of children under 7 years of age as a hetero-assessment and directly to children over 7 years of age as a selfassessment.
* Parental Stress Index - Short Form (PSI-SF): Short version of the Parental Stress Index. The instrument will be offered to parents of study participants in self-report. It evaluates the magnitude of stress in the parent-child system.

Interventions :

The study has two phases:

The clinician-led interview will be conducted with the parent(s) or directly with the child in a face-to-face or remote setting.

-The scales will be validated via an online platform. An initial analysis of the general data (primary and secondary criteria) will be carried out using various descriptive statistics indicators. Depending on the participation rate in the study and the total number of participants, a general linear model analysis will be performed on the different indicators collected (presence/absence of the different symptoms, and scores on the different instruments) in order to describe the evolution of the children's symptoms. The data collected in this study will then be compared to the initial post-exposure assessment.

Duration: The estimated duration of the study is one year (including analyses). Participation in the inclusion period is six months. The duration of participation per person in the study will be 30 minutes of interview + 20 minutes of delivery of psychological instruments.

ELIGIBILITY:
Inclusion Criteria:

* Child and/or young adult aged under 18 at the time of exposure having been assessed by the CUMPS teams during the "ALEX Storm" interventions of October 2020
* Affiliated to a social security scheme
* Children whose parents have accepted participation in the study and/or young adults who have accepted participation in the study (collection of non-objection

Exclusion Criteria:

* Children and/or young adults with a severe somatic and/or psychiatric disorder that makes assessment impossible or may alter emotional regulation behavior.
* Non-participation in a parallel study that could modify emotional regulation behavior

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children of adolescents who were seen by the teams of the Cellules d'Urgence Médico-Psychologique (CUMP) following the Alex storm in October 2020.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
diagnostic criteria for post-traumatic stress disorder | at inclusion
  Semi-structured interview based on the Clinician-Administered PTSD scale for DSM-5 Child/Adolescent -CAPS-CA-5. This instrument allows for the This instrument is validated in English, and a French translation was carried out by the investigators (translation/back-translation method). The instrument uses the DSM-5 diagnostic criteria for post-traumatic stress disorder (PTSD).
  This tool as 517 items. This scale doesn't work on numerical values (there is no min, max or cut scores), this scale makes it possible to confirm or invalidate the presence of symptoms necessary for establishing diagnoses on Diagnosis and Statistical Manual of Mental Disorders (DSMV) criteria

SECONDARY OUTCOMES:
intensity of the symptoms | at inclusion
  The intensity of the symptoms of this PTSD will be assessed by the Young Child PTSD checklist (YCPC) for young children under the age of 7. For children over 7 years of age, it will be assessed by the Child PTSD checklist, child version (CPC)
  These scales aim to screen for post-traumatic stress disorder symptoms in children aged 1 to 6 years old, by evaluating traumatic exposures (13 items), symptoms presented by the child (23 items) and his level of impairment or functional impairment (6 items). Items 14 to 36 relate to symptoms of PTSD and are based on a 5-points Likert scale, each item is scored from 0 to 4, the YCPC has a score ranging from 0 to 92. The diagnosis Cutoff is at 26 or more for items 14-36, it indicates a "probable diagnosis" of PTSD.
assessment of somatization | at inclusion
  Patient Health Questionnaire 13 items (PQH13). This simple and quick to use instrument allows a systematic assessment of somatization in children. This questionnaire will be offered to parents of children under 7 years of age as a hetero-assessment and directly to children over 7 years of age as a selfassessment
  Thirteen items, each of which is scored 0 to 2, providing a 0 to 30 severity score.
Parental Stress | at inclusion
  Parental Stress Index - Short Form (PSI-SF): Short version of the Parental Stress Index. The instrument will be offered to parents of study participants in self-report. It evaluates the magnitude of stress in the parent-child system The "Parental Stress Index Short Form" is a self-assessment intended for the child's parent The PSI-SF has 36 items from the original 120-item PSI and based on a 5-points Likert scale, each item is scored from 1 to 5, the PSI-SF has a score ranging from 36 to 180. Percentile scores are used to interpret the scores.
  Scores at or above the 85th percentile are considered high (normal range : 15th-80th percentile

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Pediatriques de Nice Chu-Lenval, Nice, France